CLINICAL TRIAL: NCT06863285
Title: The Pharmacist Led Educational Interventions Through Telemedicine to Improve Asthma Control: a Randomized Control Trial
Brief Title: Asthma Control Through Telemedicine
Acronym: PLET-I
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Muhammad Abubakar, Assistant professor, Hamdard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ABJan012025
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Asthmatic Patients
Keywords: Asthma; Telemedicine; pharmacist
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): intervention included the usual counselling by pharmacist e.g. Patients Education regarding Medications
  * Pharmacist counseling patients regarding their disease and severity
  * Pharmacist counseling (5- to 10-minute sessions) on the proper and safe use of medication.
  * Pharmacist counseling patients regarding the importance of their therapy (treatment), non-pharmacological treatment like diet and exercises.
  pharmacist counselling regarding the preventive measures that prevent patient from triggers that can initiate asthmatic attacks.
  Interventions: Other: Educational
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Educational — intervention included the usual counselling by pharmacist e.g. Patients Education regarding Medications
  * Pharmacist counseling patients regarding their disease and severity
  * Pharmacist counseling (5- to 10-minute sessions) on the proper and safe use of medication.
  * Pharmacist counseling patients regarding the importance of their therapy (treatment), non-pharmacological treatment like diet and exercises.
  pharmacist counselling regarding the preventive measures that prevent patient from triggers that can initiate asthmatic attacks.
  Arms: Study group

SUMMARY:
The purpose of this research study is to evaluate the impact of pharmacist led educational interventions on Asthmatic patients, and also determine their medication adherence.

Pharmacist's intervention aims to answer:

1. How a pharmacist intervention program impact medication adherence in persistent asthma?
2. To assess how pharmacist led educational intervention like patients' counseling and medication reminders through Telemedicine have an impact on patient's asthma control?
3. Which mode of communication (Verbal instructions, videos and pamphlets) for the patient counselling is most beneficial for the patients in asthma control.

DETAILED DESCRIPTION:
This is a randomized, pharmacist-led, two-group, longitudinal descriptive interventional study performed through in person (Public and private hospitals) and telecommunication (WhatsApp, network calls and messaging). The investigator will use snowball method to approach patients through telecommunication. Recruited patients will be randomly divided into two groups: the Control and the experimental group. The Control Group will not receive any intervention, and experimental group will receive special counseling about persistent asthma, it's medications and medical devices, their appropriate use, and side effects. Using Telemedicine as message and call reminders to increase medication adherence and improve their asthmatic condition. The intervention will be conducted for one month on the experimental group according to the recruitment date and time of the patients.

Pre-validated questionnaires will be used for the assessment

1. The adherence to asthma medication questionnaire (AAMQ-13).
2. Asthma Control test TM (ACT).

ELIGIBILITY:
Inclusion Criteria:

* Age above 11 years.
* Persistent Asthma Patient.
* Patients taking medications and inhaler.
* Patient who will consent for the study.
* Patient with basic telecommunication facility.
* Patient who responded to messages and calls.

Exclusion Criteria:

* Patients who will refuse to participate in study will not be included.
* Irresponsive patients to messages and calls

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Score | 1 month
  Patient health related outcomes that is level of asthma control is measured by pre-validated tool Asthma Control test TM (ACT).
  The Asthma Control Test™ assess responsiveness to changes in asthma control over time.
  The tool has 5 questions with each having options with scores 1,2,3,4, and 5. A SCORE OF 19 OR LESS might be a warning of the need for further evaluation to determine whether adjustments to asthma treatment regimens or other measures are required to improve asthma control. If score is 15 or less, asthma may be poorly controlled or not controlled at all.
Patients Medication Adherence Score | 1 month
  The primary aim of this study will be to evaluate the effectiveness/impact of a pharmacist educational intervention on medication adherence in Asthmatic patients.
  Adherence will be measured using the adherence to asthma medication questionnaire (AAMQ-13 The AAMQ-13 is a reliable and valid questionnaire with several desirable characteristics as it has a high internal validity, good criterion validity, and strong construct validity. The AAMQ-13 is a suitable questionnaire that can identify non-adherent patients and reveal the reasons behind their non-adherence (intentional or unintentional non-adherence). Each question has Always, Often, sometimes, rarely and never response with scores allotted as 1,2,3,4 and 5 respectively, Score interpretation is as follows for the given tool Poor adherence Score= 13-29 Moderate adherence Score= 30-47 Excellent adherence= 48-65

CONTACTS AND LOCATIONS:
Locations (1):
- Hamdard University, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The participant's identity is to be kept strictly confidential as per consent form that will be prepared for the study.